CLINICAL TRIAL: NCT04938856
Title: A Single Center, Open Label, Randomized, Single-dose, 2 Way Cross-over Study to Explore the Bioequivalence of Lamnet (Lamotrigine)100mg Tablet With the Reference Product Lamictal 100mg (Lamotrigine) Tablet Under Fasting Conditions in Healthy Male Pakistani Subjects
Brief Title: Bioequivalence of Lamnet (Lamotrigine)100mg Tablet With the Reference Product Lamictal 100mg (Lamotrigine) Tablet Under Fasting Conditions
Acronym: BE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: The Searle Company LTD., Pakistan. (Unknown)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-026-LAM-2018/Protocol/2.0
Record Dates: First submitted 2021-06-12; First posted 2021-06-24 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Bioequivalence
Keywords: Bioequivalence Study; Healthy Volunteers; Pakistani Population; Safety
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Intervention Model Description: open label, randomized, single-dose, 2 way cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Oral administration of Lamnet (100mg) Tablet after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time-point.
  Interventions: Drug: Lamotrigine tablet
- Reference Group (Active Comparator): Oral administration of Lamictal (100mg) Tablet after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time-point.
  Interventions: Drug: Lamotrigine tablet

INTERVENTIONS:
Drug: Lamotrigine tablet — Lamotrigine 100 mg immediate release Tablet
  Other Names: Test Group (Lamnet 100 mg), Reference Group (Lamictal 100 mg)

SUMMARY:
Single oral administrations of study drug (Lamnet and Lamictal) in two periods separated by a washout period of 14 days. The washout period will be calculated from day of dosing (Day 2) to at least 14 days post dose in each period.

DETAILED DESCRIPTION:
The study drugs will be administered with 240 mL ambient Temperature water after at least 10 hours fasting in each periods.

Pharmacokinetic parameters include Lamotrigine plasma concentrations at the given sampling times. In each period 18 blood samples for plasma Lamotrigine concentrations will be taken on Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7 (at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5 ,4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post-dose.) The primary parameters to be analyzed are the maximum plasma concentration (Cmax), area under the plasma concentration-time curve from zero to the time of the last measurable time point t (AUClast or also termed as AUC0-t) and area under the plasma concentration-time curve from zero to infinity (AUCtotal or, also termed as AUC0-inf) and (AUC0-t)/ (AUC0-inf).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 55 years inclusive.
* Subjects with a body mass index from 18.5 to 30 kg/m2 (both inclusive).
* Subjects who are healthy as determined by routine physical examination, including vital sign monitoring (i.e., blood pressure, heart rate and temperature), ECG monitoring and laboratory analysis (ie, hematology, blood biochemistry, and urinalysis)and viral serology as determined by the investigator.
* Tested negative for COVID-19 (through COVID-19 antibody testing).
* Subjects should have negative urine test for drugs of abuse (morphine, cannabinoids will be tested) and alcohol breath analysis at screening and prior to each check-in.
* Subjects will be able to, understand and sign the Informed Consent Form for Medical Screening during their screening visit and Participation Informed Consent Form on study check-In day.
* Subject agreed not to use special diet including fasting, high protein diet within the next 4 weeks.
* Subject agreed not to consume Alcohol, cigarette, gutka, caffeine or related xanthines containing foods or beverages (e.g. tea, coffee, cola drinks, chocolates, cocoa) etc and poppy seeds (khash khash) within 48 hours prior to drug administration.
* Subject agreed not to intake prescription drugs within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medicine.
* Subject agreed not to intake non-prescription drugs (OTC) within 14 days prior to first dose of study medicine.
* Subject agreed to discontinue vitamins ,dietary and herbal supplements within 14 days prior to the first dose of study medication.
* Subject agreed not to consume grapefruit and/or its products within 14 days prior to the start of study.

Exclusion Criteria:

* Inability to take oral medication.
* Tested positive for COVID-19 (through COVID-19 antibody testing).
* History of smoking (≤3cigarette/day), alcoholism, and positive test for drug of abuse, heavy pan or gutka user as judged by teeth / mouth inspection.
* Subjects with clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication.
* Subject is allergic to Lamotrigine and any of the product of lamotrigine .
* Subject has received any investigational drug within four weeks.
* Participated in any clinical trials within 30 days.
* Subjects with salt imbalance in the blood (especially low levels of potassium or magnesium in the blood).
* Donation or loss of more than 450 mL of blood within 3 months prior to the screening.
* History of any significant illness in the last four weeks which might confound in the result of the study or post additional risk in administrating lamotrigine to the subject.
* Concomitant treatment with Valproate, Carbamazepine, phenytoin, phenobarbital, primidone,, rifampin, Estrogen-containing oral contraceptives, Protease inhibitors lopinavir/ritonavir and atazanavir/lopinavir.
* Subjects who test positive for syphilis (VDRL) or who are known to have serum hepatitis or who are carriers of the Hepatitis B surface antigen (HBs Ag) or are carriers of antibodies to hepatitis C virus (anti-HCV) or to the human immunodeficiency virus (HIV-1 or HIV-2).
* Individuals having undergone any major surgery within 3 months prior to the start of the study, unless deemed eligible, otherwise by the Principal Investigator or whomever he/she may designate.
* Subjects with any condition, which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or elimination of drugs.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of asthma, anaphylaxis or anaphylactic reactions, severe allergic responses.
* Current or past history of nervous-psychiatric disorder, in the opinion of investigator that the subject is at risk of suicide or with history of suicide behavior/attempt.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pakistani Population
Enrollment: 26 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-120 hours post dose
  maximum plasma concentration of Lamotrigine
AUC | 0 to 120 hours post dose
  Area Under the Plasma Drug Concentration versus Time curve
Tmax | 0-120 hours post dose
  Time required for maximum plasma drug concentration

SECONDARY OUTCOMES:
Blood Pressure monitoring | 0-120 hours post dose
  monitoring if blood pressure after dose administration
Body temperature measurement | 0-120 hours post dose
  Measurement of body temprature after dose administration
Heart rate measurement | 0-120 hours post dose
  Measurement of heart rate after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad R Shah, PhD, Principal Investigator — Center for bio-equivalence studies and clinical research, ICCBS, University of Karachi; Dr. Naghma Hashmi (Co-PI), PhD, Principal Investigator — Center for bio-equivalence studies and clinical research, ICCBS, University of Karachi
Locations (1):
- Center for Bioequivalence Studies and clinical research, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The study related information can be obtained via proper request to the PI unless the confidentiality of the participants are not compromised.